CLINICAL TRIAL: NCT04484441
Title: Maternal-fetal Immune Responses to Fetal Surgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mauro H. Schenone, Principal Investigator, Mayo Clinic
Other Study IDs: 19-011382
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Spina Bifida; Congenital Diaphragmatic Hernia; Lower Urinary Tract Obstructive Syndrome; Myelomeningocele
Keywords: Fetal Surgery; Fetal Intervention; In Utero Surgery; In Utero Intervention
MeSH Terms: conditions — Spinal Dysraphism; Hernias, Diaphragmatic, Congenital; Meningomyelocele | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fetal surgical intervention group: Pregnant adult women carrying a fetus with a diagnosed congenital anomaly and scheduled to undergo fetal surgical intervention at Mayo Clinic.
  Interventions: Other: Blood and placenta specimen collection.
- Control group - normal pregnancy: Pregnant adult women with normal ultrasound findings. These women will be matched with the subjects enrolled in the intervention cohort for parity, maternal age, ethnicity, fetal sex and gestational age at time of surgical intervention.
  Interventions: Other: Blood and placenta specimen collection.

INTERVENTIONS:
Other: Blood and placenta specimen collection. — Collection of maternal and paternal blood. Collection of infant cord blood and placenta.

SUMMARY:
Performing surgery in utero on fetuses with certain birth defects has led to significant improvements in outcomes after birth; however, many of these infants are born preterm which can decrease the effectiveness of these procedures. The investigators aim to understand the effects of surgery on the maternal and fetal immune system and whether immune activation may be causing some of these infants to be born prematurely.

DETAILED DESCRIPTION:
Over 300,000 neonates worldwide die in their first month of life due to a congenital birth defect. Thanks to advancements in diagnostic technology and imaging, the field of fetal surgery was developed to treat some of these conditions in utero. Results have demonstrated improved short and long-term outcomes following surgery, especially for those fetuses diagnosed with congenital diaphragmatic hernia, lower urinary tract obstruction and spina bifida. However, over 30% of the surgical cases will have preterm labor, leading to complications related to neonatal prematurity. The cause of this surgery-induced preterm birth is unknown; however, disruption in fetal-maternal tolerance may lead to immune activation and inflammation of the maternal and fetal immune systems. Maintaining immunologic tolerance is essential during pregnancy, as a women shares only half of her genetic material with the fetus. Previous work has demonstrated that fetal surgery leads to an increase in maternal cells identified in cord blood. Animal studies have also shown that in utero intervention leads to the activation of maternal cells against fetal (paternal) antigen. Based on this previous data, it is hypothesized that surgical trauma following in utero intervention results in mixing of maternal and fetal cells leading to activation of systemic (adaptive maternal immunity) and regional (fetal placental macrophages) immune responses that disrupt fetal-maternal tolerance, which can result in preterm birth. Blood will be collected from pregnant women and their partners. Blood and placental tissue will be collected from infants that do and do not undergo in utero surgery to determine whether maternal T cells specific to fetal antigen are activated and expand after in utero intervention; and 2) to determine whether placental macrophages (Hofbauer Cells) and histology in the maternal-fetal interface exhibit increased activation and inflammation in surgical cases born preterm (<37 weeks) compared to term. Should this exploratory study reveal activation of maternal and/or fetal immune responses following in utero surgery, modalities aimed at therapeutically suppressing these acute responses may prolong gestation, significantly benefiting newborns diagnosed with a congenital anomaly.

ELIGIBILITY:
Inclusion Criteria for study group:

* Maternal age ≥18 years
* Pregnant with a congenital anomaly diagnosis AND undergoing fetal intervention in utero
* Delivery planned at Mayo Clinic, Rochester MN

Inclusion Criteria for control group:

* Maternal age ≥18 years
* Pregnant with normal ultrasound findings
* Delivery planned at Mayo Clinic, Rochester MN

Exclusion Criteria:

* Delivery planned elsewhere
* Abnormal fetal karyotype

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will compare two groups of pregnant women. Each group will be comprised of maternal, paternal, fetal trios. The study cohort will be comprised of adult women carrying a fetus with a diagnosed congenital anomaly and scheduled to undergo fetal surgical intervention. The control cohort will enroll pregnant women with normal ultrasound findings that will be matched with the subjects enrolled in the study cohort for parity, maternal age, ethnicity, fetal sex and gestational age at time of surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Maternal T cell activation following in utero intervention. | Baseline, 1-2 days post intervention, 1 week post intervention, delivery
  T cells from maternal blood will be isolated and CDR3 spectra typing will be completed. These samples will be compared to each other to identify high frequency T cell clones as well as longitudinal changes in the dynamics of clones.
  Blood collected at the four time points above will be profiled for changes in immune activation using mass cytometry (CyTOF) and plasma collected to measure changes in cytokine responses pre- and post-surgery by multiplex.

SECONDARY OUTCOMES:
Placental histology in the maternal-fetal interface in term and preterm fetal intervention cases | Delivery
  Placental macrophages will be phenotyped for subtypes (M1 classical versus M2 repair), activation (CD25 and CD40), and apoptosis status by CyTOF. Comparisons will be made between those born before 37 weeks and those born after 37 weeks in the surgical group, as well as to those who didn't undergo surgery.
  From each placenta, 5 sections will be dissected and submitted for histological evaluation of placental villitis. Toxoplasmosis, Other [syphilis, varicella-zoster, parvovirus B19], Rubella, Cytomegalovirus and Herpes (TORCH) infection panels will be completed to distinguish infectious villitis from immune-mediated villitis.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Schenone, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Texas Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials